CLINICAL TRIAL: NCT03149952
Title: A Pilot Study of the Feasibility of Setting up a Logbook for Allogeneic Haematopoietic Stem Cell Patients at the University Hospital of Amiens
Acronym: CABALLO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator choice
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2016_843_0012
Record Dates: First submitted 2017-05-02; First posted 2017-05-11 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Allogeneic Disease; Hematopoietic Stem Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient hospitalized for allogeneic haematopoietic stem cells (Other)
  Interventions: Other: Evaluation of the feasibility of the establishment of a logbook in patients hospitalized for allogeneic haematopoietic stem cells

INTERVENTIONS:
Other: Evaluation of the feasibility of the establishment of a logbook in patients hospitalized for allogeneic haematopoietic stem cells — Evaluation of the feasibility of the establishment of a logbook in patients hospitalized for allogeneic haematopoietic stem cells.

SUMMARY:
Hospitalization for allogeneic haematopoietic stem cell transplantation constitutes a particular time in the management of patients with malignant hemopathies both for the patient, for his entourage or for the nursing staff. For the patient, the strict protective isolation set up during this period is a source of isolation in the broad sense and is associated with an escape from external events and society. It also constitutes a physical barrier (mask, charlotte, surblouse and overshoes worn by caregivers or visitors) and even psychological in relations with relatives. Moreover, this period is also difficult because of the possible complications of conditioning (mucositis, transit disorders, fever ...) and allograft itself (graft versus host disease, no transplant, relapse disease…). The patient may be weakened and diminished, which can give a feeling of helplessness and uselessness to the family. Finally, this therapy can have serious physical and psychological consequences for the patient and his entourage (especially in the case of family allograft) who do not always have the possibility to express themselves verbally. Published studies in hematology report depressive, anxious and post-traumatic stress disorders in patients and relatives during allogeneic haematopoietic stem cell transplantation. It is therefore important to reduce these symptoms, particularly those related to the cut-off during hospitalization for allogeneic haematopoietic stem cells.

Over the last decade or so, the logbook has been used in some resuscitation services in intubated patients, with the main objective of filling the "memory gap" mentioned by the intubated patients when they woke up and limiting the trauma associated with this Cut in the world corresponding to the sedation period. For this purpose, the use of a logbook in Hematology, by analogy with what is used in the resuscitation services, could be a means of limiting the psychological complications related to the allograft.

ELIGIBILITY:
Inclusion Criteria:

* Major hospitalized patient for allogeneic haematopoietic stem cells
* Patient agreeing to participate

Exclusion Criteria:

* Patient refusing to participate
* Patient hospitalized for reasons other than allogeneic haematopoietic stem cells

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Analysis of the effectiveness of the logbook made available to hospitalized patients in hematology to limit the psychological complications related to the allograft. | 1 year